CLINICAL TRIAL: NCT01360086
Title: Trial Evaluating the Efficacy and Tolerance of Perioperative Chemotherapy With 5FU-Cisplatin-Cetuximab in Adenocarcinomas of the Stomach and Gastroesophageal Junction. Phase II Single Arm, Multicenter.
Brief Title: Fluorouracil, Cisplatin, Leucovorin Calcium, and Cetuximab in Treating Patients With Adenocarcinoma of the Stomach or Gastroesophageal Junction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000699219; FFCD-0901; EU-21111; EUDRACT-2010-023115-33; MERCK-FFCD-0901
Record Dates: First submitted 2011-05-20; First posted 2011-05-25 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Gastric Cancer
Keywords: adenocarcinoma of the gastroesophageal junction; adenocarcinoma of the stomach; stage IB gastric cancer; stage IIA gastric cancer; stage IIB gastric cancer; stage IIIA gastric cancer; stage IIIB gastric cancer; stage IIIC gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cetuximab; Cisplatin; Fluorouracil; Leucovorin; Chemotherapy, Adjuvant; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perioperative CT with 5FU-Cisplatine-Cetuximab (Experimental): 6 cycles of intravenous Cetuximab (500mg/m²), Cisplatine (50mg/m²) and LV5FU2s (folinic acid 400mg/m², 5FU bolus 400mg/m², and continuous infusion of 5FU 2400mg/m²) every 2 weeks. Surgery was planned 3-4 weeks after the end of neaodjuvant CT and postoperative CT, with the same regimen, planned for 6-8 weeks after surgery.
  Interventions: Biological: cetuximab; Drug: cisplatin; Drug: fluorouracil; Drug: leucovorin calcium; Procedure: adjuvant therapy; Procedure: neoadjuvant therapy; Procedure: quality-of-life assessment; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Biological: cetuximab — 6 cycles of intravenous Cetuximab (500mg/m²),
Drug: cisplatin — Cisplatine (50mg/m²)
Drug: fluorouracil — LV5FU2s (folinic acid 400mg/m², 5FU bolus 400mg/m², and continuous infusion of 5FU 2400mg/m²) every 2 weeks
Drug: leucovorin calcium
Procedure: adjuvant therapy
Procedure: neoadjuvant therapy
Procedure: quality-of-life assessment
Procedure: therapeutic conventional surgery — Surgery was planned 3-4 weeks after the end of neaodjuvant CT

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil, cisplatin, and leucovorin calcium, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving more than one drug (combination chemotherapy) together with cetuximab before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving these drugs after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying the side effects of giving fluorouracil, cisplatin, and leucovorin calcium together with cetuximab and to see how well they work in treating patients with adenocarcinoma of the stomach or gastroesophageal junction.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the objective response rate according to RECIST V1.1 criteria in patients with adenocarcinoma of the stomach or gastroesophageal junction treated with neoadjuvant chemotherapy comprising fluorouracil, cisplatin, leucovorin calcium, and cetuximab followed by surgery and adjuvant chemotherapy.
* To determine the non-toxicity rate in these patients.

Secondary

* To determine the rate of macroscopically and microscopically complete surgical resection (R0).
* To determine the overall tolerance in patients treated with this regimen.
* To determine post-operative mortality and morbidity in these patients.
* To determine the rate of recurrence at 1 and 2 years in these patients.
* To determine recurrence-free survival at 3 years in these patients.
* To determine disease-free survival at 3 years in these patients.
* To determine overall survival at 3 years in these patients.
* To determine quality of life using EORTC QLC-C30 and STO-22 questionnaires.
* To determine the correlation between the response rate and the degree of skin toxicity.

OUTLINE: This is a multicenter study.

* Neoadjuvant therapy and surgery: Patients receive leucovorin calcium IV over 2 hours, cisplatin IV, fluorouracil IV continuously over 46 hours, and cetuximab IV over 1-2 hours on day 1. Treatment repeats every 2 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Within 3-4 weeks after completing neoadjuvant chemotherapy, patients undergo surgery.
* Adjuvant therapy: Within 4-8 weeks after completing neoadjuvant chemotherapy, patients receive leucovorin calcium, cisplatin, fluorouracil, and cetuximab as in neoadjuvant therapy. Treatment repeats every 2 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients complete quality-of-life questionnaires (QLC-C30 and STO-22) periodically. Blood and tissue samples are collected periodically for correlative and translational studies.

After completing study therapy, patients are followed up every 4 months for 2 years and then every 6 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the stomach or gastroesophageal junction

  * Stage IB, II, or III disease according to TNM classification OR type I, II, or III disease according to Siewert classification

    * TNM: T1N1-3, T2N0-3, T3N0-3, or T4N0-3 (no T1N0 or M1)
  * Disease considered operable with curative intent
* No gastric scirrhous carcinoma (linitis plastica)

  * Forms with independent cells are not considered linitis
* Measurable disease according to RECIST V1.1
* No planned esophagectomy without thoracotomy in patients with adenocarcinoma of the gastroesophageal junction type I

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Polynuclear neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine clearance > 50 mL/min
* Bilirubin < 1.5 times normal
* Serum albumin > 30 g/L
* Prothrombin time ≥ 80%
* FEV1 > 1 L in case of thoracotomy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known cirrhosis
* No other progressive condition that has not been stabilized including the following:

  * Hepatic failure
  * Renal failure
  * Respiratory failure
  * NYHA class III-IV congestive heart failure
  * Unstable angina
  * Myocardial infarction in the past 6 months
  * Significant arrhythmias in the past 12 months
* No recent weight loss exceeding 15%
* No interstitial pneumonia
* No other malignant tumor within the past 5 years except for basal cell skin carcinoma or cancer in situ of the cervix
* No psychological, familial, or geographical reasons that will preclude the patient being monitored regularly
* No persons deprived of liberty or under guardianship (Disability Act)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy or radiotherapy for gastric cancer
* No other concurrent anticancer treatment, immunotherapy, or hormone therapy
* No prior abdominal or thoracic radiotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Objective response rate according to RECIST V1.1 criteria | 3 months
Non-toxicity rate | 3 months

SECONDARY OUTCOMES:
Tolerance | From Inclusion
Post-operative mortality and morbidity | After Surgery
Rate of recurrence at 1 and 2 years | 1 year and 2 years
Recurrence-free survival at 3 years | 3 years
Disease-free survival at 3 years | 3 years
Overall survival at 3 years | 3 years
Quality of life as assessed by QLC-C30 and STO-22 questionnaires | From inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Mariette, MD, PhD, Principal Investigator — Centre Hospitalier Regional et Universitaire de Lille
Locations (2):
- France (2):
  - Centre Hospitalier Regional et Universitaire de Lille, Lille
  - CHU - Robert Debre, Reims

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mariette C, Dahan L, Mornex F, Maillard E, Thomas PA, Meunier B, Boige V, Pezet D, Robb WB, Le Brun-Ly V, Bosset JF, Mabrut JY, Triboulet JP, Bedenne L, Seitz JF. Surgery alone versus chemoradiotherapy followed by surgery for stage I and II esophageal cancer: final analysis of randomized controlled phase III trial FFCD 9901. J Clin Oncol. 2014 Aug 10;32(23):2416-22. doi: 10.1200/JCO.2013.53.6532. Epub 2014 Jun 30. PMID 24982463
- [Derived] Gronnier C, Mariette C, Lepage C, Monterymard C, Jary M, Ferru A, Baconnier M, Adhoute X, Tavan D, Perrier H, Guerin-Meyer V, Lecaille C, Bonichon-Lamichhane N, Pillon D, Cojocarasu O, Egreteau J, D'journo XB, Dahan L, Locher C, Texereau P, Collet D, Michel P, Ben Abdelghani M, Guimbaud R, Muller M, Bouche O, Piessen G. Perioperative Cetuximab with Cisplatin and 5-Fluorouracil in Esogastric Adenocarcinoma: A Phase II Study. Cancers (Basel). 2023 Apr 6;15(7):2188. doi: 10.3390/cancers15072188. PMID 37046849